CLINICAL TRIAL: NCT04363164
Title: A Randomized Phase II Study Comparing Sequential High Dose Testosterone and Enzalutamide to Enzalutamide Alone in Asymptomatic Men With Castration Resistant Metastatic Prostate Cancer
Brief Title: Sequential Testosterone and Enzalutamide Prevents Unfavorable Progression
Status: Recruiting | Phase: Phase 2 | Type: Interventional
Sponsor: Sidney Kimmel Comprehensive Cancer Center at Johns Hopkins (Other)
Collaborators: United States Department of Defense (U.S. Federal Agency)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: J2060sIRB; IRB00312725 (Other: JHU IRB)
Record Dates: First submitted 2020-04-23; First posted 2020-04-27 (Actual); Last update posted 2025-07-14 (Actual); Status verified 2025-07

CONDITIONS: Castration Resistant Metastatic Prostate Cancer
Keywords: Testosterone; Enzalutamide; Androgen Deprivation Therapy (ADT)
MeSH Terms: interventions — testosterone 17 beta-cypionate; enzalutamide; testosterone enanthate

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No | US Export: No

ARMS (3):
- Arm A: Enzalutamide (Experimental): Patients randomized to Arm A will receive continuous therapy with standard dose Enzalutamide (160 mg oral daily).
  Interventions: Drug: Enzalutamide
- Arm B: Sequential Testosterone and Enzalutamide (Experimental): Patients in Arm B will receive intramuscular injection with testosterone cypionate (T) at a dose of 400 mg every 28 days x 2 (i.e. cycle 1). On Day 1 of cycle 2, patients will stop testosterone and begin enzalutamide 160 mg po q day for 56 days. Each cycle is 56 days. On Day 1 of cycle 3, patient will not take enzalutamide and will again receive injection of testosterone. Patients will continue to alternate one cycle of testosterone (2 injections) with one cycle of 56 days of enzalutamide.
  Interventions: Drug: Testosterone cypionate; Drug: Enzalutamide; Drug: Testosterone enanthate
- Arm C: Variable Sequential Testosterone and Enzalutamide (Experimental): Patients in Arm C will receive intramuscular injection with testosterone cypionate (T) at a dose of 400 mg every 28 days x 2 injections per cycle. Each cycle is 56 days. Patients with PSA progression will stop T injection and begin Enzalutamide. Patients on T with initial PSA decline will remain on high dose T for additional cycles of 2 injections until PSA progression occurs (≥25% increase in PSA from PSA nadir on current BAT cycle). These patients will then be started on Enzalutamide. Patients with PSA progression will stop Enzalutamide and will restart injections of T with 2 injections/cycle. Patients on enzalutamide with initial PSA decline after one 56-day cycle will continue on Enzalutamide until PSA progression occurs (≥25% increase in PSA from PSA nadir on current Enzalutamide cycle). These cycles of switching between T and Enza with onset of PSA progression will continue until clinical and/or radiographic progression occurs.
  Interventions: Drug: Testosterone cypionate; Drug: Enzalutamide; Drug: Testosterone enanthate

INTERVENTIONS:
Drug: Testosterone cypionate — Depo-Testosterone Injection, for intramuscular injection, contains testosterone cypionate which is the oil-soluble of the androgenic hormone testosterone. Testosterone cypionate is a white or creamy white crystalline powder, odorless or nearly so and stable in air. Depo-Testosterone Injection is available in two strengths, 100 mg/mL and 200 mg/mL testosterone cypionate.
  Other Names: Depo-Testosterone Injection
  Arms: Arm B: Sequential Testosterone and Enzalutamide; Arm C: Variable Sequential Testosterone and Enzalutamide
Drug: Enzalutamide — Enzalutamide is a white crystalline non-hygroscopic solid. It is practically insoluble in water. Enzalutamide is provided as liquid-filled soft gelatin capsules for oral administration. Each capsule contains 40 mg of enzalutamide as a solution in caprylocaproyl polyoxylglycerides. The inactive ingredients are caprylocaproyl polyoxylglycerides, butylated hydroxyanisole, butylated hydroxytoluene, gelatin, sorbitol sorbitan solution, glycerin, purified water, titanium dioxide, and black iron oxide.
Drug: Testosterone enanthate — Testosterone Enanthate Injection, for intramuscular injection, contains testosterone enanthate which is the oil-soluble ester of the androgenic hormone testosterone. Enanthate Injection is available as a colorless to pale yellow solution. Each mL contains 200 mg testosterone enanthate in sesame oil with 5 mg chlorobutanol as a preservative.
  Other Names: Delatestryl
  Arms: Arm B: Sequential Testosterone and Enzalutamide; Arm C: Variable Sequential Testosterone and Enzalutamide

SUMMARY:
Asymptomatic men without pain due to prostate cancer progressing with metastatic CRPC after treatment with combination or sequential ADT + Abi will be treated on a randomized, open label study to determine if sequential treatment with high dose T and Enza will improve primary and secondary objectives vs. continuous Enza as standard therapy.

DETAILED DESCRIPTION:
Eligible patients are those who have progressive disease after treatment with Abi either in combination with ADT as initial therapy or as second-line therapy after development of resistance to primary ADT. Patients will continue on ADT with LHRH agonist (i.e. Zoladex, Trelstar, Eligard or Lupron) or LHRH antagonist (Degarelix) if not surgically castrated throughout the duration of the study to inhibit endogenous testosterone production. Patients will be randomized 1:2:2 and stratified based on whether they received Abi in combination with ADT or in sequence after progression on ADT and based on duration of response to Abi (<6 or ≥ 6 months).

Patients randomized to Arm A will receive continuous therapy with standard dose Enza (160 mg po q day).

Patients randomized to Arm B will receive Sequential Testosterone and Enzalutamide (STE). Patients in Arm B will receive intramuscular injection with testosterone cypionate (T) at a dose of 400 mg every 28 days x 2 (i.e. cycle 1). This dose was selected based on data demonstrating that it produces an initial high dose serum level of T (i.e. > 1500 ng/dL or 3-10 times normal level) with eugonadal levels achieved at the end of two weeks and near castrate levels after 28 days. On Day 1 of cycle 2, patients will stop testosterone and begin enzalutamide 160 mg po q day for 56 days. Each cycle is 56 days. On Day 1 of cycle 3, patient will not take enzalutamide and will again receive injection of testosterone. Patients will continue to alternate one cycle of testosterone (2 injections) with one cycle of 56 days of enzalutamide.

Patients randomized to Arm C will receive Variable Sequential Testosterone and Enzalutamide (VSTE). Patients in Arm C will receive intramuscular injection with testosterone cypionate (T) at an FDA-approved dose of 400 mg every 28 days x 2 injections per cycle. Patients will remain on high dose T for at least one cycle. Each cycle is 56 days. Patients with PSA progression (≥25% increase in PSA from baseline PSA on BAT cycle) will stop T injection and begin Enzalutamide. Patients on T with initial with declining PSA decline PSA will remain on high dose T for additional cycles of 2 injections until PSA progression occurs (≥25% increase in PSA from PSA nadir on current BAT cycle)based on PCWG3 criteria. Patients with PSA progression (≥25% increase in PSA from baseline) will stop T injection. These patients will then be started on Enzalutamide. Patients with PSA progression (≥25% increase in PSA from baseline on enzalutamide cycle) will stop Enzalutamide and will restart injections of T with 2 injections/cycle. Patients on enzalutamide with initial PSA decline after one 56- day cycle will continue on Enzalutamide until PSA progression occurs (≥25% increase in PSA from PSA nadir on current Enzalutamide cycle). . Patients with PSA progression (≥25% increase in PSA from baseline) will stop Enzalutamide and will restart injections of T with 2 injections/cycle. These cycles of switching between T and Enza with onset of PSA progression will continue until clinical and/or radiographic progression occurs.

Patients will have prostate-specific antigen (PSA) level and symptoms assessment checked every cycle. Every 2 cycles (~4 months) patients will have repeat bone/CT scans to evaluate treatment response status. On CT scan, radiographic progression will be defined by RECIST criteria (i.e. >20% increase in the sum of target lesions). On bone scan, radiographic progression will be defined by PCWG3 criteria as ≥ 2 new bone lesions.

Patients with PSA progression but with disease response or stable disease on imaging studies will remain on study until clinical or radiographic progression criteria are met. Patients with radiographic disease progression will stop treatment and come off study. Patients with clinical progression due to pain flare after first two injection of testosterone can remain on study. If pain persists after first cycle of enzalutamide, patients will stop treatment and come off study. If pain resolves on enzalutamide, but returns with next or subsequent cycles of testosterone, patients will stop treatment and come off study.

ELIGIBILITY:
Inclusion Criteria:

1. ECOG Performance status ≤2.
2. Age ≥18 years.
3. Histologically-confirmed adenocarcinoma of the prostate.
4. Treated with continuous androgen ablative therapy (either surgical castration or LHRH agonist/antagonist).
5. Documented castrate level of serum testosterone (<50 ng/dl).
6. Metastatic disease radiographically documented by CT or bone scan.
7. Must have had disease progression while on combination of abiraterone acetate plus ADT either given concurrently or sequentially based on:

   * PSA progression defined as an increase in PSA, as determined by 2 separate measurements taken at least 1 week apart And/ Or
   * Radiographic disease progression, based on RECIST 1.1 in patients with measurable soft tissue lesions or PCWG3 for patients with bone disease
8. Screening PSA must be ≥ 1.0 ng/mL.
9. Patients with soft tissue lesion amenable to biopsy must agree to biopsy collection pre-treatment and at a defined point on treatment to perform tumor tissue analysis.
10. No prior treatment with enzalutamide, apalutamide, darolutamide, or other investigational AR targeted treatment is allowed.
11. Prior treatment with testosterone is allowed.
12. Prior treatment with one chemotherapy regimen with docetaxel (≤ 6 doses) for hormonesensitive prostate cancer is allowed.
13. Prior treatment with Provenge vaccine and 223Radium (Xofigo) is allowed if >4 weeks from last dose.
14. Patients must be withdrawn from abiraterone for ≥ 2 weeks.
15. Attempts must be made to wean patients off prednisone prior to starting therapy. Patients who cannot be weaned due to symptoms may continue on lowest dose of prednisone achieved during weaning period.
16. Acceptable liver function:

    1. Bilirubin < 2.5 times institutional upper limit of normal (ULN)
    2. AST (SGOT) and ALT (SGPT) < 2.5 times ULN
17. Acceptable renal function:

    a. Serum creatinine < 2.5 times ULN
18. Acceptable hematologic status:

    1. Absolute neutrophil count (ANC) ≥ 1500 cells/mm3 (1.5 ×109/L)
    2. Platelet count ≥ 100,000 platelet/mm3 (100 ×109/L)
    3. Hemoglobin ≥ 8 g/dL.
19. At least 4 weeks since prior radiation or chemotherapy.
20. Ability to understand and willingness to sign a written informed consent document.

Exclusion Criteria:

1. Pain due to metastatic prostate cancer requiring treatment intervention with pain medication.
2. ECOG Performance status ≥3
3. Prior treatment with enzalutamide is prohibited.
4. Prior chemotherapy with docetaxel or cabazitaxel for castration resistant prostate cancer is prohibited.
5. Requires urinary self-catheterization for voiding due to obstruction secondary to prostatic enlargement well documented to be due to prostate cancer or benign prostatic hyperplasia (BPH). Patients with indwelling Foley or suprapubic catheter for obstructive symptoms are eligible.
6. Evidence of disease in sites or extent that, in the opinion of the investigator, would put the patient at risk from therapy with testosterone (e.g. femoral metastases with concern over fracture risk, severe and extensive spinal metastases with concern over spinal cord compression, extensive liver metastases).
7. Evidence of serious and/or unstable pre-existing medical, psychiatric or other condition (including laboratory abnormalities) that could interfere with patient safety or provision of informed consent to participate in this study.
8. Active uncontrolled infection, including known history of HIV/AIDS or hepatitis B or C.
9. Any condition or mental impairment that may compromise the ability to give informed consent, patient's safety or compliance with study requirements as determined by the investigator.
10. Patients receiving anticoagulation therapy with warfarin, rivaroxaban, or apixaban are not eligible for study. [Patients on enoxaparin eligible for study. Patients on warfarin, rivaroxaban,or apixaban, who can be transitioned to enoxaparin prior to starting study treatments will be eligible].
11. Patients are excluded with prior history of a thromboembolic event within the last 12 months that are not being treated with systemic anticoagulation.
12. Hematocrit >51%, untreated severe obstructive sleep apnea, uncontrolled or poorly controlled heart failure [per Endocrine Society Clinical Practice Guidelines (34)]
13. Patients allergic to sesame seed oil or cottonseed oil are excluded.
14. Major surgery (eg, requiring general anesthesia) within 3 weeks before screening, or has not fully recovered from prior surgery (ie, unhealed wound). Note: subjects with planned surgical procedures to be conducted under local anesthesia may participate.

Ages: 18 Years to 90 Years | Sex: Male | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 150 (Estimated)
Dates: Start 2020-08-19 (Actual); Primary Completion 2026-07 (Estimated); Study Completion 2027-07 (Estimated)

PRIMARY OUTCOMES:
Clinical or Radiographic Progression free survival | Up to 2 years
  Time from the date of the randomization to the date of first documented radiological progression per RECIST 1.1 for soft tissue or PCWG3 for bone lesions, or clinical progression or death, whichever occurs first.

SECONDARY OUTCOMES:
Safety of cyclical parenteral testosterone as assessed by the revised National Cancer Institute Common Toxicity Criteria | Up to 2 years
  Safety of cyclical parenteral testosterone in asymptomatic men with recurrent castrate resistant prostate cancer. Safety will be evaluated by adverse events as assessed by the revised National Cancer Institute Common Toxicity Criteria (NCI CTC), version 4.0
Prostate-Specific Antigen Response Rate | Up to 2 years
  Number of participants achieving a Prostate-Specific Antigen decline ≥ 50% according to Prostate Cancer Working Group (PCWG2) criteria.
Objective Response Rate as Determined by RECIST | Up to 2 years
  Number of participants with partial (PR) or complete response (CR) as defined by response evaluation criteria in solid tumors (RECIST), where CR is a disappearance of all target lesions and PR is ≥30% reduction in the sum of the longest diameter of target lesions.
Quality of Life as Assessed by FACIT Fatigue Scale | Up to 1 year
  The Functional Assessment of Chronic Illness Therapy - Fatigue has a score range of 0-52 with higher scores indicating better quality of life.
Quality of Life as Assessed by Short Form 36 | Up to 1 year
  All questions are scored on a scale from 0 to 100. The total score from all of the questions answered is divided by the total number of the questions answered yielding a global score from 0-100 with 100 representing the highest level of functioning possible.
Time to Overall Survival | Up to 3 years
  Time to overall survival will be calculated as months from date of off treatment up to 3 years.
Radiographic Progression free survival | Up to 2 years
  Number of months until 20% increase in the sum of target lesions on CT scans or greater than 2 new bone lesions on bone scan.

CONTACTS AND LOCATIONS:
Overall Officials: Samuel Denmeade, MD, Principal Investigator — SKCCC at Johns Hopkins
Locations (6):
- United States (6):
  - University of California, San Diego (UCSD), San Diego, California
  - Johns Hopkins University/Sidney Kimmel Cancer Center, Baltimore, Maryland
  - Dana-Faber Cancer Institute, Boston, Massachusetts
  - University of Minnesota, Minneapolis, Minnesota
  - University of Nebraska Medical Center, Omaha, Nebraska
  - University of Washington/Fred Hutchinson Cancer Center, Seattle, Washington

IPD SHARING:
Plan to Share IPD: No